CLINICAL TRIAL: NCT00945893
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety of MEDI3414 in Adults
Brief Title: A Study to Evaluate the Safety of H1N1 Monovalent Vaccine (MEDI3414) in Healthy Adults
Acronym: MI-CP215
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MI-CP215; HHS/ASPR (Other Grant/Funding Number: HHSO100200900002I)
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Results first posted 2011-09-05 (Estimated); Last update posted 2011-09-12 (Estimated); Status verified 2011-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MEDI3414 [Influenza A (H1N1) vaccine] (Experimental): MEDI3414 - Monovalent vaccine was supplied in intranasal sprayers containing a total volume of 0.5mL of sucrose-phosphate buffer, egg allantoic fluid, and approximately 10^7 fluorescent focus units (FFU) of live, attenuated influenza virus reassortant A/California/7/2009 strain that was propagated in chicken eggs. H1N1 monovalent influenza vaccine (MEDI3414) contained no preservatives and no adjuvants.
  Interventions: Biological: MEDI3414 [Influenza A/H1N1 live attenuated, intranasal]
- Placebo (Placebo Comparator): Placebo -Placebo was supplied in intranasal sprayers containing 0.5 mL of sucrose-phosphate buffer.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: MEDI3414 [Influenza A/H1N1 live attenuated, intranasal] — 0.5 mL; (intranasal sprayer)
  Other Names: MEDI3414
  Arms: MEDI3414 [Influenza A (H1N1) vaccine]
Other: Placebo — (intranasal sprayers containing 0.5 mL of sucrose-phosphate buffer)
  Arms: Placebo

SUMMARY:
The purpose of this study was to determine the safety and descriptive immunogenicity of the H1N1 influenza vaccine in healthy adults.

DETAILED DESCRIPTION:
The primary objective of this study was to assess the safety and descriptive immunogenicity of a monovalent influenza virus vaccine containing a new 6:2 influenza virus reassortant in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 49 years of age (not yet reached their 50th birthday) at the time of randomization
* Healthy by medical history and physical examination
* Written informed consent and any locally required authorization (eg, Health Insurance Portability and Accountability Act [HIPAA] in the United States of America [USA], European Union [EU] Data Privacy Directive in the EU) obtained from the subject/legal representative prior to performing any protocol-related procedures, including screening evaluations
* Females of childbearing potential, (ie, unless surgically sterile [eg, bilateral tubal ligation, bilateral oophorectomy, or hysterectomy], has sterile male partner, is at least 1 year post menopause, or practices abstinence) must use an effective method of avoiding pregnancy (including oral, transdermal, or implanted contraceptives, intrauterine device, female condom with spermicide, diaphragm with spermicide, cervical cap, or use of a condom with spermicide by the sexual partner) for 30 days prior to the first dose of investigational product, and must agree to continue using such precautions for 60 days after the second dose of investigational product. In addition, the subject must also have a negative urine or blood pregnancy test at screening and, if screening and Day 1 do not occur on the same day, on the day of vaccination prior to randomization.
* Males, unless not sexually active, must use an effective method of birth control with a female partner and must agree to continue using such contraceptive precautions for at least 30 days after the second dose of investigational product (from Day 1 through Day 59 of the study)
* Subject is available by telephone
* Subject is able to understand and comply with the requirements of the protocol, as judged by the investigator
* Subject is able to complete follow-up period of 180 days after Dose 2 as required by the protocol

Exclusion Criteria:

* History of hypersensitivity to any component of the investigational product including egg or egg protein, gelatin or arginine, or serious, life-threatening, or severe reactions to previous influenza vaccinations
* History of hypersensitivity to gentamicin
* Any condition for which the inactivated influenza vaccine is indicated, including chronic disorders of the pulmonary or cardiovascular systems (eg, asthma), chronic metabolic diseases (eg, diabetes mellitus), renal dysfunction, or hemoglobinopathies that required regular medical follow-up or hospitalization during the preceding year
* Acute febrile (> 100.0°F oral or equivalent) and/or clinically significant respiratory illness (eg, cough or sore throat) within 14 days prior to randomization
* History of asthma
* Any known immunosuppressive condition or immune deficiency disease, including human immunodeficiency virus infection, or ongoing immunosuppressive therapy
* History of Guillain-Barré syndrome
* A household contact who is severely immunocompromised (eg, hematopoietic stem cell transplant recipient, during those periods in which the immunocompromised individual requires care in a protective environment); subject should additionally avoid close contact with severely immunocompromised individuals for at least 21 days after receipt of investigational product
* Receipt of any investigational agent within 30 days prior to randomization, or expected receipt through 30 days after the second dose of investigational product (use of licensed agents for indications not listed in the package insert is permitted)
* Expected receipt of antipyretic or analgesic medication on a daily or every other day basis from randomization through 14 days after receipt of each dose of investigational product
* Administration of intranasal medications within 14 days prior to randomization, or expected receipt through 14 days after administration of each dose of investigational product
* Receipt of any nonstudy vaccine within 30 days before or after Dose 1 or expected receipt of any nonstudy vaccine within 30 days before or after Dose 2
* Known or suspected mitochondrial encephalomyopathy
* Subject is pregnant or a nursing mother
* Any condition (eg, chronic cough, allergic rhinitis) that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results
* Subject or immediate family member of subject is an employee of the clinical study site or is otherwise in involved with the conduct of the study

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2009-08; Primary Completion 2009-09 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raburn Mallory, M.D., Study Director — MedImmune LLC
Locations (5):
- United States (5):
  - Covance Daytona Beach, Daytona Beach, Florida
  - Pharmax Research Clinic, Miami, Florida
  - Miami Research Associates, South Miami, Florida
  - Center for Pharmaceutical Research, Kansas City, Missouri
  - Clinical Research Associates, Inc., Nashville, Tennessee

REFERENCES:
- [Derived] Mallory RM, Malkin E, Ambrose CS, Bellamy T, Shi L, Yi T, Jones T, Kemble G, Dubovsky F. Safety and immunogenicity following administration of a live, attenuated monovalent 2009 H1N1 influenza vaccine to children and adults in two randomized controlled trials. PLoS One. 2010 Oct 29;5(10):e13755. doi: 10.1371/journal.pone.0013755. PMID 21060780

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened for the study within 14 days prior to randomization. The first and last dates of informed consent were 03 Aug 2009 and 18 Aug 2009. Once informed consent was obtained, a subject identification number was assigned using an interactive voice response system, and screening evaluations began to assess study eligibility.
Pre-assignment Details: Eligible subjects were randomly assigned in a 4:1 ratio to receive 2 doses of monovalent vaccine or placebo by intranasal spray; the doses were administered approximately 28 days apart, on Days 1 and 29.
Groups:
- Placebo: Placebo (intranasal sprayers containing 0.5 mL of sucrose-phosphate buffer). Subjects received two doses by intranasal spray administered approximately 28 days apart on Days 1 and 29.
- MEDI3414 [Influenza A (H1N1) Vaccine]: MEDI3414 - Monovalent vaccine was supplied in intranasal sprayers containing a total volume of 0.5mL of sucrose-phosphate buffer, egg allantoic fluid, and approximately 10^7 FFU (fluorescent focus units) of live, attenuated influenza virus reassortant A/California/7/2009 strain that was propagated in chicken eggs. H1N1 monovalent influenza vaccine (MEDI3414) contained no preservatives and no adjuvants.
Period: Overall Study
Arm/Group | Placebo | MEDI3414 [Influenza A (H1N1) Vaccine]
Started | 60 | 240
Day 15 Post Dose 1 | 60 | 238
Day 15 Post Dose 2 | 54 | 226
Completed | 57 | 230
Not Completed | 3 | 10
Not completed — Lost to Follow-up | 2 | 8
Not completed — Withdrawal of consent | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo (intranasal sprayers containing 0.5 mL of sucrose-phosphate buffer). Subjects received two doses by intranasal spray; each dose was administered approximately 28 days apart on Days 1 and 29.
- Total: Total of all reporting groups
Arm/Group | Placebo | MEDI3414 [Influenza A (H1N1) Vaccine] | Total
Number analyzed (Participants) | 60 | 240 | 300
Age Continuous [Mean (Standard Deviation); unit: years] | 34.1 (8.9) | 33.3 (9.2) | 33.5 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 138 | 171
  Male | 27 | 102 | 129
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 95 | 113
  Not Hispanic or Latino | 42 | 145 | 187
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Number; unit: participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 13 | 37 | 50
  White | 47 | 199 | 246
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Fever Post Dose 1 (Days 1-8), Defined as an Oral Temperature ≥ 101°F (38.3°C).
Description: The number of participants with fever between the two treatment groups was compared based on the upper limit of the two-sided 95% exact confidence intervals (CIs) for the rate difference (Vaccine minus Placebo). The upper limit of the two-sided 95% CI was evaluated against the prespecified equivalence criterion of 10% which corresponded to the following hypotheses • H0 (null): rate difference ≥ 10% • HA (alternative): rate difference < 10%
Time Frame: Days 1-8
Population: Safety Population was defined as all participants who received at least one dose of investigational product and had any follow-up for safety.
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI3414 [Influenza A (H1N1) Vaccine]
Number analyzed (Participants) | 60 | 240
Participants | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs MEDI3414 [Influenza A (H1N1) Vaccine]; The upper limit of the two-sided 95% CI was evaluated against the prespecified equivalence criterion of 10% which corresponded to the following hypotheses: H0 (null): Rate Difference ≥ 10%, HA (alternative): Rate Difference < 10%; Test type: Non-Inferiority or Equivalence — The currently proposed study provided at least 99.9% power to rule out a rate increase of 10 percentage points assuming the true difference between the treatment groups is zero and the true fever rate is ≤ 3%. Power is also high if the true difference is slightly greater than zero and the true fever rate is ≤ 3%; Score; Rate difference = 0.0, 95% CI 2-sided [-6.0 to 1.9]

2. Primary Outcome: Number of Participants Who Experienced a Post Dose 1 (Day 15) Seroresponse Against the H1N1 Strain in All Participants Regardless of Baseline Serostatus
Description: Seroresponse was defined as a ≥ 4-fold rise in hemagglutination inhibition (HAI) titer from baseline. All immunogenicity analyses were based on the immunogenicity population.
Time Frame: Day 1, Day 15
Population: For each treatment group, participants were randomized at a 1:1 ratio to have their post Dose 1 immunogenicity blood draw occur on either Day 15 or Day 29. Participants who received Dose 1 of the investigational product and had valid HAI measurements from blood samples obtained at baseline and post Dose 1 were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI3414 [Influenza A (H1N1) Vaccine]
Number analyzed (Participants) | 30 | 120
Participants | 0 | 3
Statistical Analysis 1: Comparison: Placebo vs MEDI3414 [Influenza A (H1N1) Vaccine]; The number of participants who experienced a post-dose seroresponse was compared based on the upper limit of the limit of the two-sided 95% exact CI for the rate difference (Vaccine minus Placebo); Test type: Superiority or Other; score; rate difference = 2.5, 95% CI 2-sided [-8.8 to 7.7]

3. Primary Outcome: Number of Participants Who Experienced a Post Dose 1 (Day 29) Seroresponse Against the H1N1 Strain in All Participants Regardless of Baseline Serostatus
Description: Seroresponse was defined as a ≥ 4-fold rise in HAI titer from baseline. All immunogenicity analyses were based on the immunogenicity population.
Time Frame: Day 1, Day 29
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI3414 [Influenza A (H1N1) Vaccine]
Number analyzed (Participants) | 29 | 115
Participants | 0 | 7
Statistical Analysis 1: Comparison: Placebo vs MEDI3414 [Influenza A (H1N1) Vaccine]; The number of participants who experienced a post-dose seroresponse was compared based on the upper limit of the two-sided 95% exact CIs for the rate difference (Vaccine minus Placebo); Test type: Superiority or Other; score; rate difference = 6.1, 95% CI 2-sided [-5.6 to 12.6]

4. Primary Outcome: Number of Participants Who Experienced a Post Dose 2 (Day 57) Seroresponse Against the H1N1 Strain in All Participants Regardless of Baseline Serostatus
Description: as for outcome 3
Time Frame: Day 1, Day 57
Population: Participants who received 2 doses of the same investigational product and had valid HAI measurements from blood samples obtained at baseline and post Dose 2 were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI3414 [Influenza A (H1N1) Vaccine]
Number analyzed (Participants) | 54 | 222
Participants | 3 | 33
Statistical Analysis 1: Comparison: Placebo vs MEDI3414 [Influenza A (H1N1) Vaccine]; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; score; rate difference = 9.3, 95% CI 2-sided [-0.8 to 16.3]

5. Secondary Outcome: Number of Participants With Any Solicited Symptom Within 7 Days Post Vaccination, Dose 1
Description: Solicited symptoms were events considered likely to occur post dosing. For this study, other solicited symptoms included: Fever (> 100°F [37.8°C] oral), Runny nose, Sore throat, Cough, Vomiting, Muscle aches, Chills, Decreased activity (tiredness), and Headache.
Time Frame: Days 1-8
Population: The Safety population for solicited symptoms was defined as all participants who received at least one dose of investigational product, had any follow-up for safety and had solicited symptom data available during the reporting period.
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI3414 [Influenza A (H1N1) Vaccine]
Number analyzed (Participants) | 60 | 240
Participants | 19 | 100
Statistical Analysis 1: Comparison: Placebo vs MEDI3414 [Influenza A (H1N1) Vaccine]; Test type: Non-Inferiority or Equivalence — Rates of solicited symptoms following each dose (Days 1 to 8 and Days 1 to 15) between the two treatment groups were compared following each dose. Exact two-sided 95% CIs (Chan and Zhang, 1999) on the rate difference (monovalent vaccine minus placebo) were constructed. There were no prespecified equivalence criteria for the secondary analyses; Score; Rate difference = 10.0, 95% CI 2-sided [-4.1 to 22.8]

6. Secondary Outcome: Number of Participants Reporting Adverse Events (AEs) Within 7 Days Post Vaccination, Dose 1
Time Frame: Days 1-8
Population: The Safety Population was defined as all participants who received at least one dose of investigational product and had any follow-up for safety.
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI3414 [Influenza A (H1N1) Vaccine]
Number analyzed (Participants) | 60 | 240
Participants | 7 | 26

7. Secondary Outcome: Number of Participants Using Anti-pyretic and Analgesic Agents Within 7 Days Post Vaccination, Dose 1.
Time Frame: Days 1-8
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI3414 [Influenza A (H1N1) Vaccine]
Number analyzed (Participants) | 60 | 240
Participants | 3 | 20

8. Secondary Outcome: Number of Participants With Any Solicited Symptom Within 14 Days Post Vaccination, Dose 1
Time Frame: Days 1-15
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI3414 [Influenza A (H1N1) Vaccine]
Number analyzed (Participants) | 60 | 240
Participants | 28 | 113
Statistical Analysis 1: Comparison: Placebo vs MEDI3414 [Influenza A (H1N1) Vaccine]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Score; Rate difference = 0.4, 95% CI 2-sided [-13.9 to 14.5]

9. Secondary Outcome: Number of Participants Reporting AEs Within 14 Days Post Vaccination, Dose 1
Time Frame: Days 1-15
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI3414 [Influenza A (H1N1) Vaccine]
Number analyzed (Participants) | 60 | 240
Participants | 10 | 38

10. Secondary Outcome: Number of Participant Using Anti-pyretic and Analgesic Agents Within 14 Days Post Vaccination, Dose 1
Time Frame: Days 1-15
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI3414 [Influenza A (H1N1) Vaccine]
Number analyzed (Participants) | 60 | 240
Participants | 3 | 30

11. Secondary Outcome: Number of Participants With Any Solicited Symptom Within 7 Days Post Vaccination, Dose 2
Time Frame: Days 29-36
Population: The Safety Population for solicited symptoms dose 2 was defined as all participants who received Dose 2, had any follow-up for safety and had solicited symptom data available during the reporting period.
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI3414 [Influenza A (H1N1) Vaccine]
Number analyzed (Participants) | 55 | 228
Participants | 15 | 61
Statistical Analysis 1: Comparison: Placebo vs MEDI3414 [Influenza A (H1N1) Vaccine]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Score; Rate difference = -0.5, 95% CI 2-sided [-14.7 to 11.8]

12. Secondary Outcome: Number of Participants Reporting AEs Within 7 Days Post Vaccination, Dose 2
Time Frame: Days 29-36
Population: Participants in the Safety Population who received Dose 2 and had any follow-up for safety during the reporting period.
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI3414 [Influenza A (H1N1) Vaccine]
Number analyzed (Participants) | 55 | 228
Participants | 3 | 12

13. Secondary Outcome: Number of Participants Using Anti-pyretic and Analgesic Agents Within 7 Days Post Vaccination, Dose 2
Time Frame: Days 29-36
Population: Participants in the safety population who received Dose 2 and had any follow-up for safety during the reporting period.
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI3414 [Influenza A (H1N1) Vaccine]
Number analyzed (Participants) | 55 | 228
Participants | 2 | 4

14. Secondary Outcome: Number of Participants With Any Solicited Symptom Within 14 Days Post Vaccination, Dose 2
Time Frame: Days 29-43
Population: Participants in the Safety Population who received Dose 2 and had solicited symptom data available during the reporting period.
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI3414 [Influenza A (H1N1) Vaccine]
Number analyzed (Participants) | 55 | 228
Participants | 17 | 75
Statistical Analysis 1: Comparison: Placebo vs MEDI3414 [Influenza A (H1N1) Vaccine]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Score; Rate difference = 2.0, 95% CI 2-sided [-12.6 to 14.9]

15. Secondary Outcome: Number of Participants Reporting AEs Within 14 Days Post Vaccination, Dose 2
Time Frame: Days 29-43
Population: Participants in the Safety Population who received Dose 2 and had any follow-up for safety during the reporting period.
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI3414 [Influenza A (H1N1) Vaccine]
Number analyzed (Participants) | 55 | 228
Participants | 4 | 18

16. Secondary Outcome: Number of Participants Using Anti-pyretic and Analgesic Agents Within 14 Days Post Vaccination, Dose 2
Time Frame: Days 29-43
Population: Participants in the Safety Population who received Dose 2 and had any follow-up for safety during the reporting period.
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI3414 [Influenza A (H1N1) Vaccine]
Number analyzed (Participants) | 55 | 228
Participants | 2 | 10

17. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) Through 28 Days Post Vaccination, Dose 1
Description: SAEs were those AEs that resulted in death; were immediately life threatening; resulted in inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability or incapacity; were a birth defect in the offspring of a participant; or were an important medical event that may not have resulted in death, threatened life, or required hospitalization and that, based on appropriate medical judgment, may have jeopardized the participant and may have required medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: Days 1-29
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI3414 [Influenza A (H1N1) Vaccine]
Number analyzed (Participants) | 60 | 240
Participants | 0 | 0

18. Secondary Outcome: Number of Participants With New Onset Chronic Diseases (NOCDs) Within 28 Days Post Vaccination, Dose 1
Description: An NOCD was a newly diagnosed medical condition that was of a chronic, ongoing nature and was assessed by the investigator as medically significant. Examples of NOCDs included, but were not limited to, diabetes, asthma, autoimmune disease (eg, lupus, rheumatoid arthritis), and neurological disease (eg, epilepsy, autism). Examples of events not considered NOCDs were mild eczema, diagnosis of a congenital anomaly present at study entry, or acute illness (eg, otitis media, bronchitis).
Time Frame: Days 1-29
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI3414 [Influenza A (H1N1) Vaccine]
Number analyzed (Participants) | 60 | 240
Participants | 0 | 1

19. Secondary Outcome: Number of Participants With SAEs Through 28 Days Post Vaccination, Dose 2
Description: as for outcome 17
Time Frame: Days 29-57
Population: Participants in the Safety Population for Dose 2 who received Dose 2 and had any follow-up for safety during the reporting period.
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI3414 [Influenza A (H1N1) Vaccine]
Number analyzed (Participants) | 55 | 228
Participants | 0 | 0

20. Secondary Outcome: Number of Participants With NOCDs Within 28 Days Post Vaccination, Dose 2
Description: as for outcome 18
Time Frame: Days 29-57
Population: Participants in the Safety Population for Dose 2 who received Dose 2 and had any safety follow-up during the reporting period.
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI3414 [Influenza A (H1N1) Vaccine]
Number analyzed (Participants) | 55 | 228
Participants | 0 | 0

21. Secondary Outcome: Number of Participants With SAEs Through 180 Days Post Final Dose
Description: as for outcome 17
Time Frame: Days 1-209
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI3414 [Influenza A (H1N1) Vaccine]
Number analyzed (Participants) | 60 | 240
Participants | 2 | 3

22. Secondary Outcome: Number of Participants With NOCDs Through 180 Days Post Final Dose.
Description: as for outcome 18
Time Frame: Days 1-209
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI3414 [Influenza A (H1N1) Vaccine]
Number analyzed (Participants) | 60 | 240
Participants | 1 | 1

23. Secondary Outcome: Number of Participants Who Achieved a Post Dose 1 (Day 15) HAI Titer ≥ 32 Against the H1N1 Strain in All Participants Regardless of Baseline Serostatus
Description: All immunogenicity analyses are based on the immunogenicity population.
Time Frame: Day 1, Day 15
Population: Participants were randomized at a 1:1 ratio to have their post Dose 1 immunogenicity blood draw on either Day 15 or Day 29. Participants who received Dose 1 of the investigational product and had valid HAI measurements from blood samples obtained at baseline and post Dose 1 were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI3414 [Influenza A (H1N1) Vaccine]
Number analyzed (Participants) | 30 | 120
Participants | 1 | 11
Statistical Analysis 1: Comparison: Placebo vs MEDI3414 [Influenza A (H1N1) Vaccine]; The number of participants who achieved a post Dose 1 HAI titer greater than or equal to 32 against the H1N1 strain was compared based on the upper limit of the two-sided 95% exact CI for the rate difference (Vaccine minus Placebo); Test type: Superiority or Other; score; rate difference = 5.8, 95% CI 2-sided [-7.7 to 13.8]

24. Secondary Outcome: Number of Participants Who Achieved a Post Dose 1 (Day 29) HAI Titer ≥ 32 Against the H1N1 Strain in All Subjects Regardless of Baseline Serostatus
Description: All immunogenicity analyses are based on the immunogenicity population.
Time Frame: Day 1, Day 29
Population: as for outcome 23
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI3414 [Influenza A (H1N1) Vaccine]
Number analyzed (Participants) | 29 | 115
Participants | 4 | 9
Statistical Analysis 1: Comparison: Placebo vs MEDI3414 [Influenza A (H1N1) Vaccine]; [analysis description as in outcome 23, analysis 1]; Test type: Superiority or Other; score; rate difference = -6.0, 95% CI 2-sided [-23.5 to 5.3]

25. Secondary Outcome: Number of Participants Who Achieved a Post Dose 2 (Day 57) HAI Titer ≥ 32 Against the H1N1 Strain in All Participants Regardless of Baseline Serostatus
Description: All immunogenicity analyses are based on the immunogenicity population.
Time Frame: Day 1, Day 57
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI3414 [Influenza A (H1N1) Vaccine]
Number analyzed (Participants) | 54 | 222
Participants | 6 | 30
Statistical Analysis 1: Comparison: Placebo vs MEDI3414 [Influenza A (H1N1) Vaccine]; The number of participants who achieved a post Dose 2 HAI titer greater than or equal to 32 against the H1N1 strain was compared based on the upper limit of the two-sided 95% exact CI for the rate difference (Vaccine minus Placebo); Test type: Superiority or Other; score; rate difference = 2.4, 95% CI 2-sided [-9.3 to 10.8]

26. Secondary Outcome: Serum HAI Geometric Mean Titers (GMTs) in All Participants Regardless of Baseline Serostatus, Dose 1 (Day 15)
Description: All immunogenicity analyses are based on the immunogenicity population.
Time Frame: Day 1, Day 15
Population: as for outcome 23
Measure: Geometric Mean (Full Range); unit: Titer
Arm/Group | Placebo | MEDI3414 [Influenza A (H1N1) Vaccine]
Number analyzed (Participants) | 30 | 120
Titer | 2.64 [2 to 32] | 3.46 [2 to 256]

27. Secondary Outcome: Serum HAI GMTs in All Participants Regardless of Baseline Serostatus, Dose 1 (Day 29)
Description: All immunogenicity analyses are based on the immunogenicity population.
Time Frame: Day 1, Day 29
Population: as for outcome 23
Measure: Geometric Mean (Full Range); unit: Titer
Arm/Group | Placebo | MEDI3414 [Influenza A (H1N1) Vaccine]
Number analyzed (Participants) | 29 | 115
Titer | 4.96 [2 to 512] | 3.44 [2 to 128]

28. Secondary Outcome: Serum HAI GMTs in All Participants Regardless of Baseline Serostatus, Dose 2 (Day 29)
Description: All immunogenicity analyses are based on the immunogenicity population.
Time Frame: Day 1, Day 57
Population: as for outcome 4
Measure: Geometric Mean (Full Range); unit: Titer
Arm/Group | Placebo | MEDI3414 [Influenza A (H1N1) Vaccine]
Number analyzed (Participants) | 54 | 222
Titer | 3.90 [2 to 512] | 4.86 [2 to 1024]

ADVERSE EVENTS:
Time Frame: Safety evaluation consisted of AEs through 7 days and 14 days after each vaccination, SAEs and NOCDs through 28 days after each vaccination, and SAEs and NOCDs through 180 days after the final vaccination.
Description: Telephone contacts were made by site personnel to the subject at various times during the study to assess safety.
Groups:
- H1N1 Monovalent Vaccine Days 1-15; H1N1 Monovalent Vaccine Days 29-57; H1N1 Monovalent Days 58-209: A/California/7/2009 strain of the live, attenuated influenza virus reassortant 10^7 FFU that was propagated in chicken eggs. MEDI3414 contained no preservatives and no adjuvants. Subjects received two doses by intranasal spray; each dose was administered approximately 28 days apart on Days 1 and 29.
- Placebo Days 1-15; Placebo Days 29-57; Placebo Days 58-209: Placebo (intranasal sprayers containing 0.5 mL of sucrose-phosphate buffer). Subjects received two doses by intranasal spray; each dose was administered approximately 28 days apart on Days 1 and 29.
Arm/Group | H1N1 Monovalent Vaccine Days 1-15 | Placebo Days 1-15 | H1N1 Monovalent Vaccine Days 29-57 | Placebo Days 29-57 | H1N1 Monovalent Days 58-209 | Placebo Days 58-209
Serious Adverse Events (participants affected / at risk) | 0/240 | 0/60 | 0/228 | 0/55 | 3/240 | 2/60
Other Adverse Events (participants affected / at risk) | 17/240 | 9/60 | 13/228 | 1/55 | 0/240 | 0/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | H1N1 Monovalent Vaccine Days 1-15 (N=240) | Placebo Days 1-15 (N=60) | H1N1 Monovalent Vaccine Days 29-57 (N=228) | Placebo Days 29-57 (N=55) | H1N1 Monovalent Days 58-209 (N=240) | Placebo Days 58-209 (N=60)
Gallbladder disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | H1N1 Monovalent Vaccine Days 1-15 (N=240) | Placebo Days 1-15 (N=60) | H1N1 Monovalent Vaccine Days 29-57 (N=228) | Placebo Days 29-57 (N=55) | H1N1 Monovalent Days 58-209 (N=240) | Placebo Days 58-209 (N=60)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.